CLINICAL TRIAL: NCT04044547
Title: A Randomized, Double-blinded, Multiple Ascending Dose Study in Patients With Early-stage Parkinson's Disease to Evaluate the Pharmacokinetics and Safety of LY03003 Following Intramuscular Injections
Brief Title: A Study of LY03003 in Patients With Early-stage Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Beijing Bozhiyin T&S Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03003/CT-CHN-102
Record Dates: First submitted 2019-07-30; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; LY03003
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- LY03003 (Experimental)
  Interventions: Drug: Rotigotine, extended-release microspheres
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo, extended-release microspheres

INTERVENTIONS:
Drug: Rotigotine, extended-release microspheres — Four stable dose levels of LY03003 at 14, 28, 42 and 56 mg will be evaluated. For each dose level, the stable dose will be administered once a week for consecutive 5 weeks. To improve patient's tolerability, dose upward titration will be applied to 28, 42 and 56 mg dose groups according to the following schedule:
  * Patients to be enrolled to 14 mg dose group will receive 14 mg for 5 consecutive weeks.
  * Patients to be enrolled to 28 mg dose group will receive 14 mg in the first week and then 28 mg in the next 5 weeks.
  * Patients to be enrolled to 42 mg dose group will receive 14 mg in the first week, 28 mg in the second week and then 42 mg in the next 5 weeks.
  * Patients to be enrolled to 56 mg dose group will receive 14 mg in the first week, 28 mg in the second week, 42 mg in the third week and then 56 mg in the next 5 weeks.
  Arms: LY03003
Drug: Placebo, extended-release microspheres — Four stable dose levels of placebo at 14, 28, 42 and 56 mg will be evaluated. For each dose level, the stable dose will be administered once a week for consecutive 5 weeks. To improve patient's tolerability, dose upward titration will be applied to 28, 42 and 56 mg dose groups according to the following schedule:
  * Patients to be enrolled to 14 mg dose group will receive 14 mg for 5 consecutive weeks.
  * Patients to be enrolled to 28 mg dose group will receive 14 mg in the first week and then 28 mg in the next 5 weeks.
  * Patients to be enrolled to 42 mg dose group will receive 14 mg in the first week, 28 mg in the second week and then 42 mg in the next 5 weeks.
  * Patients to be enrolled to 56 mg dose group will receive 14 mg in the first week, 28 mg in the second week, 42 mg in the third week and then 56 mg in the next 5 weeks.
  Arms: Placebo

SUMMARY:
This study is to characterize the pharmacokinetics and to evaluate the safety as well as tolerability of LY03003 following multiple escalating intramuscular injections

ELIGIBILITY:
Inclusion Criteria:

* Patient had Parkinson's Disease that meet the clinical diagnostic criteria of the brain bank of the Parkinson's Disease Association of the United Kingdom.
* Patient was Hoehn & Yahr stage ≤3 (excluding stage 0) ;
* Patient was male or female aged 18 to 75 years;
* Patient had a Mini Mental State Examination (MMSE) score of ≥25;
* Patient had a Unified Parkinson's Disease Rating Scale (UPDRS) motor score (Part III) of ≤30 at Screening.
* Patient who signed the informed consent form volunteered to participate in this clinical trial and could cooperate with the prescribed inspections.

Exclusion Criteria:

* Patient had a history of pallidotomy, thalamotomy, deep brain stimulation, or fetal tissue transplant;
* Patient had dementia, schizophrenia or hallucinations, or clinically significant depression;
* Patient had a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or presence of suicidal tendency in the past year;
* Patient had a history of orthostatic hypotension.
* Patient had received therapy with a dopamine (DA) agonist either concurrently or had done so within 28 days prior to the Screening;
* Patient had received therapy with 1 of the following drugs either concurrently or within 28 days prior to Screening: monoamine oxidase B (MAO-B) inhibitors (e.g., pargyline, selegiline), DA releasing agents (e.g., amphetamine), reserpine, DA-antagonists (e.g., metoclopramide), neuroleptics, or other medications that may interact with DA function;
* Patient was currently (at the time of Screening) receiving central nervous system active therapy (e.g., sedatives, hypnotics, antidepressants, anxiolytics), unless the dose had been stable for at least 28 days prior to Screening Visit and was likely to remain stable for the duration of the study;
* Patient had a current diagnosis of epilepsy, had a history of seizures as an adult within 1 year prior to Screening, had a history of stroke or transient ischemic attack within 3 months prior to Screening;
* Patient had a history of known intolerance/hypersensitivity to non-dopaminergic antiemetics, such as domperidone, ondansetron, tropisetron;
* Patient had any other clinically relevant hepatic, renal, and cardiac dysfunction, or laboratory abnormality, which would have, in the judgment of the Investigator, interfered with the patient's ability to participate in the study;
* Patient had a history of allergic to any medication;
* Heavy smoker, alcoholic, drug addict;
* Female patients who were pregnant or were breastfeeding or were of childbearing potential without adequate contraception;
* Patient who was inappropriate to participant in the study in the judgment of the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11-22 (Actual); Primary Completion 2014-02-26 (Actual); Study Completion 2015-06-11 (Actual)

PRIMARY OUTCOMES:
LY03003 concentration in plasma | Days 1, 2, 4, 6, 8, 15, 22, 29, 30, 32, 34, 36, 38, 40, 43, and day 50

SECONDARY OUTCOMES:
Frequency of adverse events | From screening up to day 50
  Adverse events to evaluate the safety and tolerability of LY03003
Change from baseline to the end of the treatment period in the Unified Parkinson's Disease Rating Scale (UPDRS) part (Ⅲ) Total Score | screening, baseline and day 29 and Day 50
  The Unified Parkinson´s Disease Rating Scale Part Ⅲ is an accepted and validated scale for the assessment of motor function in Parkinson´s disease. Each of the 27 sub-items in the UPDRS III is measured on a scale of 0 to 4, where 0 is normal and 4 represents severe abnormalities. The total scores therefore ranges from 0 (Best score possible) to 108 (Worst score possible).